CLINICAL TRIAL: NCT06470581
Title: Clinical Effect of Thoracic Sympathetic Ganglion Block With Botulinum Toxin Type A in Patients With Upper Extremity Complex Regional Pain Syndrome: A Prospective Randomized, Double-blind, and Comparative Clinical Trial
Brief Title: Thoracic Sympathetic Ganglion Block With Botulinum Toxin Type A
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University (Other)
Responsible Party: Principal Investigator, Jeeyoun Moon, Professor, Seoul National University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2402-117-1516
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Complex Regional Pain Syndromes
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local anesthetics (Active Comparator): Total volume of 0.375% ropivacaine 3 mL will be injected in phase 2.
  Interventions: Drug: Botulinum toxin A
- Botulinum toxin A (Experimental): Total volume of BTX-A 75U in normal saline 3ml will be injected in phase 2.
  Interventions: Drug: Botulinum toxin A

INTERVENTIONS:
Drug: Botulinum toxin A — Patients were assigned 1:1 to a control group using only local anesthetics (Group A) and a BTX-A group (Group B). In Phase 1, the needle is inserted near the vertebrae T3 under fluoroscopic guidance. An 1 ml of non-ionized contrast medium is injected to evaluate the diffusion pattern, and 3ml of 0.75% ropivacaine is injected. After identifying a temperature increase in the ipsilateral palm within 20 min in the operating room with the prone position, 3 ml of 0.375% ropivacaine and botulinum toxin type A 75 IU mixed with 3 ml of non-preserved saline solution are injected in the patients in the control and botulinum toxin groups, respectively.

SUMMARY:
Thoracic sympathetic ganglion block is a percutaneous procedure that paralyzes the action of sympathetic nerves transiently by injecting a local anesthetic around the ganglion. It is performed to diagnose and treat sympathetically maintained pain in phantom limb pain or complex reginal pain syndrome patient. The temperature of the affected arm is often lower than that of the opposite side. As a result of the procedure, the patient may experience sympathetic pain relief, such as coldness, stinging, numbness of the upper extremity. If the procedure does not last long, repetitive block or chemical neurolysis or radiofrequency thermocoagulation for the sympathetic ganglion is performed.

However, even though in rare cases, chemical neurolysis is known to cause permanent plexus injury radiofrequency thermocoagulation is known to be less successful than chemical neurolysis because it is difficult to identify and stimulate the exact location of the ganglion. Therefore, it is expected that there will be a benefit to the patients if there is a procedure with long-lasting and avoiding injury.

Recently, it has been reported that botulinum toxin (BTX) has been successfully used for the treatment of pain disorders. BTX plays a role with blocking the secretion of acetylcholine from the cholinergic nerve endings. Therefore, the use of BTX is expected to prolong the effect of neural blockade because pre-ganglia sympathetic nerves are cholinergic. It is also known that the action of BTX is not permanent and BTX does not exhibit cytotoxicity or neurotoxicity. Therefore, Botulinum toxin type A (BTA) is recommended for the treatment of migraine, myofascial pain syndrome, and neuropathic pain accompanied by allodynia. This study would like show whether thoracic sympathetic ganglion block using BTA has a longer duration than conventional local anesthesia by using prospective randomized, double-blind, parallel group, and comparative clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. aged 19-80 years
2. Diagnosed with a complex regional pain syndrome (type 1 or 2) in unilateral upper extremity
3. 11-point numerical-rating-scale (NRS) pain score of 4 or higher in upper extremity
4. Temperature increase at diagnostic thoracic sympathetic ganglion block
5. Patients taking medication stably (without change in dosage/recipe) for more than 4 weeks prior to administration

Exclusion Criteria:

1. Refusal of the patient
2. Vascular disease at upper extremity
3. previous thoracic sympathetic neurolysis (thermocoagulation, chemical neurolysis)
4. coagulopathy
5. systemic infection or local infection at thoracic puncture site
6. significant deformity at thoracic spine
7. neoplasm
8. known allergic reaction with amide type local anesthetics
9. cognitive dysfunction (not understanding of numerical-rating-scale)
10. known allergic reaction with botulinum toxin
11. pregnant or feeding women
12. If the patient has participated in another clinical trial within 30 days before screening, or if passed no longer than 5-fold half-life of the clinical trial drug of the participating clinical trial

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-04-25 (Estimated); Study Completion 2027-04-25 (Estimated)

PRIMARY OUTCOMES:
The changes in average pain intensity in 4weeks | 4 weeks after procedure
  Comparison between groups of the average change in 11-point numerical rating scale pain score (0 = no pain, 10 = maximum pain imaginable) over the past 24 hours

SECONDARY OUTCOMES:
The changes in average pain intensity in 12weeks | 12 weeks after procedure
  Comparison between groups of the average change in 11-point numerical rating scale pain score (0 = no pain, 10 = maximum pain imaginable) over the past 24 hours
The changes in maximum pain intensity | 4 and 12 weeks after procedure
  Comparison between groups of the mamimum change in 11-point numerical rating scale pain score (0 = no pain, 10 = maximum pain imaginable) over the past 24 hours
The changes in pain related to procedure | 30 minutes after the procedure
  Inter- and intra-group comparison of the change in procedure-related 11-point numerical rating scale pain score (0 = no pain, 10 = maximum pain imaginable)
The change in the temperature difference | 30 minutes, 4 and 12 weeks after the procedure
  the change in the relative temperature difference on the blocked palm compared with the contralateral palm
Blood flow velosity | 30 minutes, 4 and 12 weeks after the procedure
  Comparison between groups of blood flow velosity at brachial artery using ultrasound
Korean CISS (Cold Intolerance Symptom Severity) Questionnaire | 4 and 12 weeks after the procedure
  Inter- and intra-group comparison of the change in Korean CISS score from 4 to 100 (mild, 4-25; moderate, 26-50; severe, 51-75; and extremely severe, 76-100)
Paindetect questionare (PD-Q) | 4 and 12 weeks after the procedure
  Inter- and intra-group comparison of the change in PD-Q score from 0 to 38 (total scores of less than 12 considered to represent nociceptive pain, 13-18 possible NeP, and >19 representing >90% likelihood of NeP)
Patient satisfaction | after procedure
  Patient satisfaction related to procedure using 5-pointed Likert scale (Very satisfied, Satisfied, Neither satisfied nor dissatisfied, Dissatisfied, and Very dissatisfied)
Medication change (Opioids) | 4 and 12 weeks after the procedure
  Comparison between groups of change with Morphine Equivalent Daily Dose (MEDD)
Additional intervention | 4 and 12 weeks after the procedure
  Comparison between groups of total number of additional executed sympathetic blocks